CLINICAL TRIAL: NCT00806455
Title: Exercise-Induced Bronchospasm in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, John Mastronarde, MD, John Mastronard M.D., Ohio State University
Other Study IDs: 2007H0319
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Cystic Fibrosis; Bronchospasm
Keywords: to determine how often exercise-induced bronchospasm; occurs in cystic fibrosis; Exercise-induced bronchospasm in cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis; Bronchial Spasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, sputum
Oversight: Data Monitoring Committee: No

SUMMARY:
Exercise is an important clinical feature in cystic fibrosis. Better exercise capacity has been associated with better patient outcomes and quality of life. Exercise-induced bronchospasm is a condition, often associated with asthma, which may make exercise difficult. The role that exercise-induced bronchospasm has in people with cystic fibrosis is unknown. This study is designed to determine how often exercise-induced bronchospasm occurs in cystic fibrosis.

DETAILED DESCRIPTION:
We anticipate that Visit 1 will take approximately three hours. This will include obtaining informed consent, completing baseline demographic and quality of life questionnaires, brief physical exam, measuring exhaled nitric oxide level, skin allergy testing, obtaining blood and sputum samples, and performing pulmonary function testing before and after bronchodilators.

Visit 2 will take approximately two and one-half hours. This will include performing Eucapnic Voluntary Hyperventilation, measuring exhaled nitric oxide levels, and obtaining blood and sputum samples.

Visit 3 will take approximately two and one-half hours. This will include performing Cardiopulmonary exercise testing followed by serial spirometry, measuring exhaled nitric oxide levels, and obtaining blood and sputum samples.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with confirmed diagnosis of Cystic Fibrosis:

   * 2 positive sweat chloride tests (or)
   * genetic testing
2. Age 12 years and older
3. Baseline FEV1 ≥70% predicted
4. Clinically stable over past 28 days:

   * no change in chronic respiratory symptoms
   * no need for antibiotics other then chronic maintenance therapies
   * no need for oral steroids
   * no increased use of bronchodilators
5. Visit 1 FEV1 within 10% of baseline

Exclusion Criteria:

1. History of Allergic Bronchopulmonary Aspergillosis (ABPA)
2. Chronic airway colonization with Burkholderia cepacia (defined as 2 or more prior positive sputum or BAL cultures)
3. Pregnancy
4. Chronic oral corticosteroid use
5. Febrile illness within two weeks of Visit 1
6. Unable to provide consent (patients under age of 18 will require both parental consent AND patient assent)
7. Current cigarette smoking, cessation of smoking within 6 weeks of Visit 1, or more than 10 pack-years of prior smoking

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Forty patients with cystic fibrosis and mild lung disease (defined by FEV1≥ 70% predicted), age 12 years and older, are our target enrollments.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of exercise-induced bronchospasm in a cohort of adolescent and adult patients with cystic fibrosis | end of study

SECONDARY OUTCOMES:
To determine the prevalence of exercise-induced bronchospasm in those CF patients with evidence of allergic inflammation versus those without allergic inflammation. | end of study
To determine the difference in exhaled nitric oxide and other surrogate markers of inflammation, as well as self-reported quality-of-life and symptom scores in CF patients with and without exercise-induced bronchospasm. | end of study

CONTACTS AND LOCATIONS:
Overall Officials: John G. Mastronarde, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Kirkby SE, Hayes D Jr, Parsons JP, Wisely CE, Kopp B, McCoy KS, Mastronarde JG. Eucapnic Voluntary Hyperventilation to Detect Exercise-Induced Bronchoconstriction in Cystic Fibrosis. Lung. 2015 Oct;193(5):733-8. doi: 10.1007/s00408-015-9745-3. Epub 2015 Jun 3. PMID 26036953